CLINICAL TRIAL: NCT00453843
Title: The Effect of Proximal and Distal Training on Stroke Recovery
Brief Title: Shoulder, or Elbow, or Wrist: What Should we Train First After a Stroke?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Burke Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD045343 (NIH)
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2007-03

CONDITIONS: Stroke
Keywords: Stroke; movement therapy; robotics; rehabilitation robotics; shoulder, elbow, wrist
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- proximal to distal training (Experimental)
  Interventions: Device: rehabilitation robotics; Procedure: Movement therapy
- distal to proximal (Experimental)
  Interventions: Device: rehabilitation robotics; Procedure: Movement therapy
- proximal and distal on alternate days (Experimental)
  Interventions: Device: rehabilitation robotics; Procedure: Movement therapy
- proximal and distal same day (Experimental)
  Interventions: Device: rehabilitation robotics; Procedure: Movement therapy

INTERVENTIONS:
Device: rehabilitation robotics — sequence of intervention
  Other Names: InMotion2.0 (InMotion Arm) and InMotion3.0 (InMotion Wrist)
Procedure: Movement therapy — sequence of intervention
  Other Names: InMotion2.0 (InMotion Arm) and InMotion3.0 (InMotion Wrist)

SUMMARY:
We will test on persons with chronic impairment due to stroke:

1. whether the order in which robot therapy is delivered influences outcomes (shoulder-and-elbow before wrist vs. wrist before shoulder-and-elbow).
2. whether we should train the shoulder, elbow, and wrist at the same time or on different days.

DETAILED DESCRIPTION:
The Effect of Proximal and Distal Training on Stroke Recovery:

Specific Aim 1. Test whether task specific wrist robotic training improves motor performance among persons with chronic impairment after stroke.

Specific Aim 2. Test whether the order in which robot therapy is delivered influences outcomes (shoulder-and-elbow before wrist vs. wrist before shoulder-and-elbow).

Specific Aim 3. Test whether there is generalization across different joints (shoulder & elbow vs wrist).

Specific Aim 4: Test whether there is any interference between training across different joints among persons with chronic impairment after stroke.

Briefly we will invite persons with chronic impairment due to stroke to participate in a study that will train them first on wrist for 6 weeks and then on the shoulder-and-elbow for an additional 6 weeks or vice-versa. A third group will train in alternate days for 12 weeks on the shoulder-and-elbow or the wrist, while a fourth group will be trained on the shoulder, elbow, and wrist on the same day. Outcomes will be measured using standard instruments as well as robot-based measures. We expect that results from this study will provide an objective basis for maximizing this kind of therapy.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the study if they meet the following criteria:

1. naïve subjects who have never experienced robot-assisted therapy as inpatients or outpatients;
2. first single focal unilateral lesion with diagnosis verified by brain imaging (MRI or CT scans) that has occurred at least 6 months prior;
3. cognitive function sufficient to understand the experiments and follow instructions (Mini-Mental Status Score of 22 and higher or interview for aphasic subjects);
4. average Motor Power score >= 1/5 or <= 3/5 (neither hemiplegic nor fully recovered motor function in 6 muscles of the shoulder, elbow, and wrist);
5. informed written consent to participate in the study.

Exclusion Criteria:

Patients will be excluded from the study if they have a fixed contraction deformity in the affected limb.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2004-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer | 3 times at baseline, midpoint, completion intervention, and at follow-up
Motor Power | 3 times at baseline, midpoint, completion intervention, and at follow-up

SECONDARY OUTCOMES:
Wolf Motor Function | 3 times at baseline, midpoint, completion intervention, and at follow-up
SIS | 3 times at baseline, midpoint, completion intervention, and at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hermano I Krebs, PhD, Principal Investigator — Massachusetts Institute of Technology
Locations (1):
- Burke Medical Research Institute, White Plains, New York, United States